CLINICAL TRIAL: NCT03571438
Title: Evaluation of a Promising New Combination of Protein Kinase Inhibitors on Organotypic Cultures of Human Renal Tumors
Acronym: COMBOREIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC17.063
Record Dates: First submitted 2018-06-15; First posted 2018-06-27 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Sunitinib; pazopanib; temsirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CK2(CX4945) and ATM(Ku 60019) (Experimental): Treatment of cell culture with a combination of CK2 and ATM inhibitors serine/ threonin Kinase combination
  Interventions: Combination Product: CK2 and ATM inhibitors serine/ threonin Kinase combination
- Sunitinib (Active Comparator): Treatment of cell culture with Sunitinib
  Interventions: Drug: Sunitinib
- Pazopanib (Active Comparator): Treatment of cell culture with Pazopanib
  Interventions: Drug: Pazopanib
- Temsirolimus (Active Comparator): Treatment of cell culture with Temsirolimus
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Combination Product: CK2 and ATM inhibitors serine/ threonin Kinase combination — Treatment of cell culture with CK2 and ATM inhibitors serine/ threonin Kinase combination
  Arms: CK2(CX4945) and ATM(Ku 60019)
Drug: Sunitinib — Treatment of cell culture with Sunitinib
  Arms: Sunitinib
Drug: Pazopanib — Treatment of cell culture with Pazopanib
  Arms: Pazopanib
Drug: Temsirolimus — Treatment of cell culture with Temsirolimus
  Arms: Temsirolimus

SUMMARY:
The investigators objective is to test the combination directly on organotypic cultures of tumors from patients after their excision in the Department of Urology and Renal Transplantation of the University Hospital of Grenoble and to compare their efficacy with that of currently selected treatments in the clinic.

The population targeted by the combination for use in clinical practice is patients with metastatic clear cell renal cell carcinoma.

Current treatments for these patients are Sunitinib, Pazopanib and Temsirolimus.

DETAILED DESCRIPTION:
Given the failure of conventional therapies in kidney cancer, both chemo and radio resistant, it was necessary to seek therapeutic alternatives.

Thus, in 2005, the first targeted therapies in kidney cancer came with protein kinase inhibitors including mTOR (mammilian target of rapamycin) inhibitors (Temsirolimus and Everolimus) and VEGFR inhibitors (Sunitinib, Sorafenib, Pazopanib and Axitinib).

Nevertheless resistance to these treatments appeared with their prolonged use as monotherapy in all cases. One of the main mechanisms of this therapeutic escape is the adaptation of the tumor cell via the use of an alternative pathway of deregulation of cell signaling.

Thus emerged the idea of simultaneously treating multiple targets to prevent the tumor cell from adapting. Phase I / II therapeutic trials have already been initiated with the combination of anti-BRAF (proto-oncogene B-Raf) and anti-MEK (MAP-ERK kinase) in metastatic melanoma or with the combination of anti-EGFR (epidermal growth factor receptor) and anti-MET in lung and breast cancer. The results are very promising since we observe a synergistic effect of two targeted therapies combined.

In kidney cancer, this escape phenomenon is also observed (example of the mTORC2 (mammilian target of rapamycin complex 2) crosstalk on AKT which limits the effect of mTORC1 (mammilian target of rapamycin complex 1) inhibitors at the level of the PI3 kinase signaling pathway).

It is therefore time to check if this strategy is applicable in kidney cancer. The investigators have, through a chemo-genomic screening of a hundred molecules stored in the CEA (French Alternative Energies and Atomic Energy Commission) chemical bank, found a combination of inhibitors targeting the kinases CK2 and ATM very effective on a human cell line of renal cell carcinoma clear. This combination has been tested on conventional cultures as well as on more innovative 3D cultures, better reproducing the tumor environment. The preliminary results obtained show that the combination is clearly more efficient in a 3D model as well as on the VHL-line (von Hippel-Lindau) in hypoxic condition, which is very encouraging.

In the context of preclinical validation, it is now essential to evaluate the therapeutic potential of these molecules by comparing their efficiency with those currently selected.

ELIGIBILITY:
Inclusion Criteria:

* major patient treated at the University Hospital of Grenoble for a renal tumor with suspected or confirmed malignancy.This includes non-metastatic patients undergoing renal lumpectomy, partial nephrectomy or total nephrectomy, as well as metastatic or locally advanced cancer patients undergoing cytoreductive surgery who are eligible for medical treatment at the same time

Exclusion Criteria:

* Contaminated patients with HIV and /or HBV (hepatitis B virus) and / or HCV (hepatitis C virus) positive serology.
* Absence or withdrawal of the informed consent of the patient.
* Tumors smaller than 2 cm on preoperative imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-16 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of cell death on organotypic cultures of human renal tumors (Efficacy) | after the treatment period (between 48 and 96 hours)
  Death cell rate on organotypic cultures of human renal tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble Alps Hospital, Grenoble, France